CLINICAL TRIAL: NCT00154154
Title: Hope for the Chronically Suicidal Patient: Evaluating the Clinical and Health Services Impact of Dialectical Behaviour Therapy in Individuals With Borderline Personality Disorder
Brief Title: Hope for the Chronically Suicidal Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Shelley McMain, Head, Borderline Personality Disorder Clinic, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIHR: #200204MCT-101123; CIHR: #200204MCT-101123
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Borderline Personality Disorder
Keywords: borderline personality disorder; BPD; treatment; dialectical behavior therapy; DBT; general Psychiatric management; GPM; suicide; parasuicide; randomized control trials
MeSH Terms: conditions — Borderline Personality Disorder; Suicide; Suicide, Attempted | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): General Psychiatric Management
  Interventions: Behavioral: General Psychiatric Management
- 2 (Experimental): Dialectal Behaviour Therapy
  Interventions: Behavioral: Dialectical Behaviour Therapy

INTERVENTIONS:
Behavioral: General Psychiatric Management — General Psychiatric Management (GPM) condition consisting of a structured algorithmic medication intervention plus psychosocial counseling.
  Arms: A
Behavioral: Dialectical Behaviour Therapy — Modification of behaviours achieved with reframing thoughts and impulses
  Arms: 2

SUMMARY:
The aim of this study is to evaluate the clinical and cost effectiveness of Dialectical Behavior Therapy (DBT) for chronically suicidal behavior in individuals diagnosed with borderline personality disorder (BPD). Recent investigations of DBT have yielded positive results and have challenged the widely held opinion that the prognosis for this condition is poor. This study will consist of a two-arm randomized controlled trial that will compare DBT with a General Psychiatric Management (GPM) condition consisting of a structured algorithmic medication intervention plus psychosocial counseling. One-hundred and eighty participants will be randomly assigned to either DBT or to the GPM condition. Clinical outcomes will be assessed by changes in: (1) parasuicidal behaviour; (2) treatment retention; (3) psychiatric symptomatology; (4) anger expression; (5) social functioning and (6) health status. Cost outcomes will include an analysis of health service utilization. Clinical and cost evaluations will occur at 4-month intervals over the course of the one-year treatment and over a two-year follow-up.

DETAILED DESCRIPTION:
Suicide, a major cause of death worldwide, is a serious public health problem. Forty percent of individuals who commit suicide meet diagnostic criteria for a personality disorder and an even higher percent of those attempting suicide have a personality disorder . Borderline personality disorder (BPD) is highly associated with parasuicidal behaviour. Parasuicidal behaviour refers to suicide attempts or other self-injurious behaviour and is a risk factor for completed suicide. Approximately 69% - 80% of people diagnosed with BPD have committed at least one act of self-harm. Estimates of completed suicides in this population are about 9%, with this rate quadrupling for patients who meet 8 or more of the 9 DSM criteria for BPD.

Chronically suicidal behaviour in people with BPD is estimated to be among the most expensive psychiatric disorders to treat. While there is an extensive anecdotal literature on the treatment of this population, clinical outcomes have been dismal and treatment evidence based on well-designed trials is sparse. Dialectical Behavior Therapy (DBT), a broad-based cognitive-behavioral therapy (CBT), has recently shown promise in the treatment of this population. DBT is being widely adopted in the treatment of this disorder despite its limited empirical base. To date, there are few studies on DBT and no replications of the original research on DBT by researchers independent of the treatment developer.

The aim of this study is to evaluate the clinical and cost effectiveness of DBT for the treatment of parasuicidal individuals with BPD compared to a General Psychiatric Management (GPM) control condition involving a structured algorithm medication intervention plus psychosocial support. This study will compare the following outcome measures in participants who receive Dialectical Behavior Therapy versus General Psychiatric Management, Best Practices during a one-year treatment interval and two-year follow-up: (1) frequency and severity of parasuicidal behaviours ; (2) number of self-harm episodes (3) improvement in quality of life (4) cost effectiveness.

Hypotheses:(1) Patients in the DBT condition will show greater reductions in the frequency and severity of parasuicidal behaviours compared to patients in the GPM condition during a one-year treatment interval and two-year follow-up; (2) Compared to GPM, DBT will result in a greater reduction in the number of self-harm episodes and a greater improvement in quality of life but will have a higher direct cost. However, because DBT will result in significant offsetting reductions in other health service costs, the incremental cost-effectiveness ratios will fall within the range of many accepted medical interventions.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV criteria for BPD
* Between 18-60 years of age
* Have had two parasuicide episodes in the past five years with one occurring in the past 3 months
* Have had OHIP coverage for 1 year or more
* Literate in English
* Provide informed consent to participate in the study

Exclusion Criteria:

* Current active substance dependence disorder
* Psychotic disorder,bipolar I disorder, or dementia
* Evidence of an organic brain syndrome or mental retardation
* A chronic or serious physical health problem that will require hospitalization within the next year (e.g. cancer)
* A medical condition that would preclude the psychiatric medication regimen in the GPM condition
* Definite plans to leave the province in the next 2 years
* Currently engaged in DBT or GPM at St. Michael's Hospital

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2002-10; Primary Completion 2007-06 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Parasuicidal behaviour | intermittent

SECONDARY OUTCOMES:
Psychiatric hospitalization | intermittent
Psychiatric symptoms | intermittent
Treatment retention | intermittent

CONTACTS AND LOCATIONS:
Overall Officials: Shelley F. McMain, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (2):
- Canada (2):
  - St Michael's Hospital, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

REFERENCES:
- [Background] American Psychiatric Association (2001). Diagnostic and Statistical Manual of Mental Disorders. Washington DC: American Psychiatric Association.
- [Background] American Psychiatric Association Practice Guidelines. Practice guideline for the treatment of patients with borderline personality disorder. American Psychiatric Association. Am J Psychiatry. 2001 Oct;158(10 Suppl):1-52. No abstract available. PMID 11665545
- [Background] Clarkin JF, Widiger TA, Frances A, Hurt SW, Gilmore M. Prototypic typology and the borderline personality disorder. J Abnorm Psychol. 1983 Aug;92(3):263-75. doi: 10.1037//0021-843x.92.3.263. No abstract available. PMID 6619404
- [Background] Cowdry RW, Pickar D, Davies R. Symptoms and EEG findings in the borderline syndrome. Int J Psychiatry Med. 1985-1986;15(3):201-11. doi: 10.2190/3y0c-hauk-04jx-gbpn. PMID 4066162
- [Background] Gunderson, J.G. (1984) Borderline Personality Disorder. Washington DC: American Psychiatric Press.
- [Background] Linehan,M.M. (1993). Cognitive-Behavorial Treatment of Borderline Personality Disorder. New York: The Guilford Press.
- [Background] Linehan, M.M. (1981). A social-behavioral analysis of suicide and parasuicide: Implications for clinical assessment and treatment. In H. Glazer & J.F. Clarkin (Eds.),Depression: Behavioral and Directive Intervention Strategies (pp. 29-294). New York: Garland.
- [Background] Linehan,MM., Heard, HL (1999). Borderline personality disorder: costs, course and treatment outcomes. In N. Mille & K. Magruder (Eds.), The cost-effectiveness of psychotherapy: Guide for practitioners, researchers and policy makers. New York: Oxford University Press, pp.291-305.
- [Background] Moscicki, E.K. (1999). Epidemiology of Suicide. In D.G. Jacobs (Ed)., The Harvard Medical School Guide to Suicde Assessment and Intervention. Josssey-Bass Publishers: San Francisco
- [Background] Paris J, Brown R, Nowlis D. Long-term follow-up of borderline patients in a general hospital. Compr Psychiatry. 1987 Nov-Dec;28(6):530-5. doi: 10.1016/0010-440x(87)90019-8. No abstract available. PMID 3691077
- [Background] Scheel,K. The empirical basis of dialectical behavioral therapy: Summary, critique and implications. Clinical Psychology-Science and Practice,2000, 7, 68-86.
- [Background] Stone, H.H. (1989). The course of borderlne personality disorder. In A. Tasman, T.E. Hales, & A.J. Frances (Eds.), American Psychiatric Press Review of Psychiatry, 8, (pp.103-122). Washington DC:American Psychiatric Press
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Runarsdottir V, Hansdottir I, Tyrfingsson T, Einarsson M, Dugosh K, Royer-Malvestuto C, Pettinati H, Khalsa J, Woody GE. Extended-Release Injectable Naltrexone (XR-NTX) With Intensive Psychosocial Therapy for Amphetamine-Dependent Persons Seeking Treatment: A Placebo-Controlled Trial. J Addict Med. 2017 May/Jun;11(3):197-204. doi: 10.1097/ADM.0000000000000297. PMID 28379861
- [Derived] McMain SF, Guimond T, Streiner DL, Cardish RJ, Links PS. Dialectical behavior therapy compared with general psychiatric management for borderline personality disorder: clinical outcomes and functioning over a 2-year follow-up. Am J Psychiatry. 2012 Jun;169(6):650-61. doi: 10.1176/appi.ajp.2012.11091416. PMID 22581157
- [Derived] McMain SF, Links PS, Gnam WH, Guimond T, Cardish RJ, Korman L, Streiner DL. A randomized trial of dialectical behavior therapy versus general psychiatric management for borderline personality disorder. Am J Psychiatry. 2009 Dec;166(12):1365-74. doi: 10.1176/appi.ajp.2009.09010039. Epub 2009 Sep 15. PMID 19755574
- See also: Web page for the Centre for Addiction and Mental Health — http://WWW.camh.net